CLINICAL TRIAL: NCT01015417
Title: Antibiotic Treatment Versus no Antibiotics in the Postoperative Acute Cholecystitis Low and Moderately Severe
Brief Title: Place of Antibiotics in the Postoperative Acute Lithiasic Cholecystitis
Acronym: ABCAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRCN09-PR-REGIMBEAU; Eudract N°2009-013470-41 (Other: AFSSAPS)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Lithiasic Cholecystitis Grade I or II; Symptoms Lasting for Less Than 5 Days; Required Cholecystectomy; Preoperative Amoxicillin Clavulanic Acid for at Most 5 Days
Keywords: Acute lithiasic cholecystitis; Cholecystectomy; Postoperative antibiotherapy; Surgical site infection; Remote surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin clavulanic acid (Active Comparator): Postoperative administration of 2g of Augmentin, 3 times daily for 5 days.
  Interventions: Drug: Amoxicillin clavulanic acid
- No medication (Other): no postoperative antibiotics
  Interventions: Other: No medication

INTERVENTIONS:
Drug: Amoxicillin clavulanic acid — Postoperative administration of 2g, 3 times daily, since 5 days, of amoxicillin clavulanic acid (Augmentin or generic) oral form or parenteral form according to clinical patient and by the choice of medical teams
  Other Names: Augmentin; generic of amoxicillin clavulanic of any brand name; ATC class J01CR02
  Arms: Amoxicillin clavulanic acid
Other: No medication — no postoperative antibiotics
  Other Names: No other name
  Arms: No medication

SUMMARY:
Assess whether postoperative antibiotics after cholecystectomy for acute lithiasic cholecystitis little or moderately severe, is effective and therefore justified.

The main objective is to compare the occurrence of postoperative infectious complications including surgical site infections (SSI) and remote infections after early cholecystectomy (performed within 5 days after onset of symptoms) for acute lithiasic cholecystitis (ALC) little or moderately serious (without organ dysfunction) with and without postoperative antibiotics.

The secondary objectives are:

* Rates of infectious complications according to duration of preoperative antibiotic
* Influence of surgical drainage after surgery for occurrence of postoperative infectious complications
* Analysis of the nature of infectious complications (surgical site infections, remote surgical site infections)
* Comparison of germs found in the bile during the postoperative infectious complications
* Duration of hospitalization
* Readmission rate for surgical site infections
* Rate of reoperation for surgical site infection
* Overall mortality rate at 30 days
* Mortality rates specific to 30 days

DETAILED DESCRIPTION:
This is a multicentre national, comparative, randomized, uncontrolled, non-inferiority, unblinded (open). Two groups of patients are compared (postoperative antibiotics versus no antibiotics postoperatively) in a ratio (1:1), intention to treat.

The international consensus conference held in Tokyo, has defined precisely the ALC(acute lithiasic cholecystis)and distinguished several stages of severity. For this study, this definition of degrees of severity will be used.

ALC is defined by the association of local signs:

* Murphy's sign
* mass
* pain
* defense of the right upper quadrant
* systemic signs (fever, leukocytosis, elevated C-reactive protein).

When the diagnosis of ALC is clinically suspected, an imaging procedure (ultrasound, a CT or MRI) is needed to confirm the diagnosis.

The morphological evidence for the diagnosis of ALC are:

* thickened gallbladder wall (> 4 mm)
* gallbladder distention (> 8cm by 4cm long axis and minor axis)
* presence of stones or debris bile (sludge)
* infiltration of fat perivesicular
* presence of an effusion perivesicular.

In this work, early ALC was defined by a disease duration of symptoms less than 5 days. This period is defined by the early onset of abdominal pain and / or fever. These criteria will be collected in case report forms.

Because the events of the ALC may range from a mild disease and confined to the gallbladder disease, to a fulminant life-threatening, a new classification of the severity of ALC has been established.

This classification has 3 levels:

* ALC mild,
* ALC moderately severe
* ALC severe.
* ALC mild (Grade I) ALC mild (Grade I) corresponds to a ALC in a patient in good general condition, without organ dysfunction, with mild inflammatory signs. At this stage there are no criteria higher stages (Grade II and III).
* ALC moderately severe (Grade II)

ALC moderately severe comprises at least one of the following criteria:

* Leukocytosis greater than 18,000 leucocytes/mm3
* Tense palpable mass on clinical examination at the right hypochondrium
* Duration of symptoms exceeding 72 hours
* Presence of local signs of inflammation (biliary peritonitis, perivesicular abscess, liver abscess, gangrenous cholecystitis, emphysematous cholecystitis)
* ALC severe (Grade III) (non-inclusion criteria of the study ABCAL)

ALC(Grade III) is accompanied by dysfunction of one of the following:

* Dysfunction Cardiovascular: hypotension requiring treatment with dopamine ≥ 5μg/kg per minute or whatever dobutamine dose.
* Neurological dysfunction: alteration of consciousness
* Respiratory dysfunction: report PaO2/FiO2 <300
* Renal dysfunction: oliguria, creatinine> 176μmol / l
* Hepatocellular dysfunction: INR> 1.5
* Hematologic dysfunction: platelet count <100 000/mm3

Patients will be included age and suffering from:

* acute lithiasic cholecystitis confirmed by morphological examination
* low and moderately severe (confined to the gallbladder)
* requiring early cholecystectomy (progression of symptoms <5 days)
* signed consent for participation

The patient will be informed of the existence of the protocol during the consultation asking the indication of cholecystectomy for acute cholecystitis.

The medical examination and imaging procedure prior to the study correspond to a routine practice (no additional cost):

A clinical examination with collection of demographic data (gender, age, weight, size) will be noted. All co-morbidities as well as situations of potential risk of infection (diabetes type 2 steroids ongoing chronic renal failure, body mass index above 30, age over 65 years, recent surgery, serum albumin less than 35 , chronic obstructive bronchitis, tobacco weaned or unweaned? coronary insufficiency) will be noted (CRF).

A review of imaging vesicular confirming the diagnosis of acute cholecystitis, which may be based on habits and ultrasound or CT and / or MRI.

All patients then selecting checking the inclusion criteria and non-inclusion will be offered to participate in the study. They will be orally informed of the progress of the study and the various examinations, an information form will be issued.

The day of surgery, after a period of reflection varies with the date and result of surgery, the inclusion visit will be conducted and include:

* The verification of inclusion criteria and non-inclusion
* A clinical examination
* The organization's planning examinations specific to the study. When the inclusion of a patient, the investigator will inform the proponent of a fax that inclusion by submitting the Form of Inclusion form (see report forms).

Patient monitoring

* Preoperative support Preoperative prescription of antibiotics will be systematic when the patient will be included in the study. The preoperative antibiotic association include: amoxicillin-clavulanate (Augmentin ® 2gx3/jour or generic with dosage equivalent). In case of allergy to beta-lactam antibiotics, the patient will be excluded from the study. Patients will be included in the study, either before hospitalization (through the use of emergency shelter), either when the patient will be hospitalized in a department (gastroenterology, geriatrics, internal medicine, etc..). A proportion of patients will have already started antibiotics (prescribed by the physician, or by the department where the patient is hospitalized). The history of antibiotics received by patients will be collected in case report forms and analyzed. For these patients, after inclusion in the study and prior cholecystectomy, antibiotic being arrested and will be replaced by amoxicillin - clavulanic acid at a dose of 2gx3/jour, in the absence of beta-lactam antibiotics allergies . The total duration of preoperative antibiotic will depend on the time of surgery and should last, in all cases, less than 5 days (inclusion criteria). The total duration of antibiotic therapy by amoxicillin - clavulanate is analyzed.
* Postoperative support The intraoperative antibiotics will be identical to the antibiotic started in preoperative(amoxicillin and clavulanic acid).

A skin preparation before surgery (antiseptic shower) and surgical (debridement and antisepsis of the operative field) will be performed. The intervention will begin with a thorough exploration of the entire peritoneal cavity and gallbladder to confirm the macroscopic diagnosis of CAL. The treatment consists of cholecystectomy with complete choice of surgical approach is left to the discretion of the operator. The laparoscopic route is preferred. The realization of a systematic sampling biliary be to compare the germs found in the gallbladder and any germs found in postoperative complications. The achievement of intraoperative cholangiography will be left to the discretion of the surgical team. The need for surgical drainage (aspiration or not) will be left to local conditions and customs of the service. The operating time will be recorded and analyzed. These variables will be collected for statistical analysis (CRF).

In the waning of the intervention, patients with bile peritonitis and those with stones in the bile duct discovered on intraoperative cholangiography can not be included in the study.

* Randomization

Randomization will be performed in the operating theater immediately after surgery. The randomization will be done by drawing lots at the patient's statement via the Internet. It will be stratified by center and to ensure a better balance, blocks of equal size with as many patients randomized to either treatment, will be used at each center.

* Postoperative management - Monitoring Visits
* Choice of postoperative antibiotic Prescription or not postoperative antibiotic, will be determined by randomization. Before administration of the antibiotic, the patients included will be questioned on the existence of a possible allergy to beta-lactam antibiotics (CRF). The postoperative antibiotic therapy will be identical to the preoperative antibiotic therapy and include the following antibiotics: amoxicillin - clavulanate (Augmentin ® 2gx3/jour). Antibiotic treatment will be issued by pharmacies centers investigators.

The combination of a nitro-imidazole is not allowed in this study. The route of administration (intravenous or oral) and the date of the relay orally depend on the clinical and biological postoperative patient are collected in case report forms. The introduction of the antibiotic will be performed in hospitals with surveillance of tolerance to the drug.

The duration of postoperative antibiotic treatment will be 5 days.

* Support during postoperative hospitalization Patients will be clinically monitored daily by the surgical team. All patients have a blood test with a blood count the day after the operation (CRF). Other blood tests may be performed according to clinical and biological patient evolution. Patients may leave the service when the surgeon deems necessary, from the 2nd postoperative day. The antibiotic treatment Augmentin ® is issued by the pharmacy at each center investigator. Antibiotics will be stored and dispensed by pharmacies in each center. Antibiotics will be issued to the patient (1 gram packets) at its output for the entire duration of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Acute lithiasic cholecystitis low or moderately severe (confined to the gall bladder)
* Requiring early cholecystectomy (progression of symptoms <5 days
* In an adult patient (>18 years)
* For each patient included the consent form must have been read, understood and signed.

Exclusion Criteria:

* Severe acute cholecystitis (with organ dysfunction)
* Acalculous cholecystitis
* Biliary peritonitis
* Abscess perivesicular
* Cholangitis
* Acute Pancreatitis
* Septic shock
* Stone of bile duct
* Physical or mental state does not allow participation in the study
* Contraindication to surgery
* Classification ASA (American Society of Anesthesiologists) IV-V or life expectancy <48 hours
* Suspected pre-or intraoperative cancer of the gallbladder
* Pregnancy or breastfeeding
* Treatment course with methotrexate, imidazole
* Known history of allergy to Augmentin ®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
All complications occurring during hospitalization or within 30 days postoperative. There are 2 main types of postoperative infectious complications: - Surgical site infections (SSI) - Systemic infections - Remote surgical site infections. | 30 days postoperative

SECONDARY OUTCOMES:
Rates of infectious complications according to duration of preoperative antibiotic | 30 days postoperative
Influence of surgical drainage after surgery for occurrence of postoperative infectious complications | 30 days postoperative
Nature of infectious complications analysis (surgical site infections, infections distance) | 30 days postoperative
Comparison of germs found in bile, the germs found in postoperative infectious complications | since the infectious complication persist
Duration of hospitalization | until the release of hospitalization, otherwise at 30 days postoperative
Readmission rate for surgical site infections (SSI) | 30 days postoperative
Rate of reoperation for SSI | 30 days postoperative
Overall mortality rate | 30 days postoperative
Specific mortality rates | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jean-marc REGIMBEAU, Pr, Study Director — Centre Hospitalier Universitaire, Amiens; David FUKS, Dr, Principal Investigator — Centre Hospitalier Universiatire Amiens
Locations (21):
- France (21):
  - Centre de Chirurgie Viscérale et de Transplantation Centre Hospitalier Régional Universitaire, Strasbourg, Alsace
  - Centre Hospitalier Haut-Lévêque, Bordeaux, Aquitaine
  - Centre Hopitalier Général, Grenoble, Auvergne-Rhône-Alpes
  - Service de Chirurgie Générale et Digestive. Centre Hospitalier Universitaire, Clermont-Ferrand, Auvergne
  - Centre Hospitalier Côte e Nacre, Caen, Basse Normandie
  - Service de Chirurgie Digestive et Vasculaire. Centre Hopsitalier Universitaire, Besançon, Doubs
  - Centre Hospitalier C.H.A.M., Rang-du-Fliers, Hauts-de-France
  - Service de Chirurgie Digetsive Centre Hopsitalier Universitaire, Montpellier, Hérault
  - Centre Hospitalier, Longjumeau, Ile de Rance
  - Centre Hospitalier Dupuytren, Limoges, Limousin
  - Chirurgie viscérale et urologique Centre Hospitalier, Beauvais, Oise
  - Centre hospitalier Universitaire, Angers, Pays de la Loire Region
  - Service de Chirurgie Viscérale et Digestive, Amiens, Picardie
  - Centre Hospitalier Timone, Marseille, Province-Alpes Côte d'Azur
  - Chirurgie Viscérale et Digestive, Rouen, Seine Maritime
  - Centre Hospitalier Jean-Verdier, Bondy, Île-de-France Region
  - Centre Hospitalier Louis Mourier, Colombes, Île-de-France Region
  - Service de Chirurgie Digestive et Viscérale, Paris, Île-de-France Region
  - Centre hospitalier Lariboisière, Paris, Île-de-France Region
  - Centre Hospitalier Cochin, Paris, Île-de-France Region
  - Centre Hospitalier de Saint-Germain en Laye, Poissy, Île-de-France Region

REFERENCES:
- [Background] Kanafani ZA, Khalife N, Kanj SS, Araj GF, Khalifeh M, Sharara AI. Antibiotic use in acute cholecystitis: practice patterns in the absence of evidence-based guidelines. J Infect. 2005 Aug;51(2):128-34. doi: 10.1016/j.jinf.2004.11.007. Epub 2005 Jan 20. PMID 16038763
- [Background] Lewis RT, Allan CM, Goodall RG, Marien B, Park M, Lloyd-Smith W, Wiegand FM. A single preoperative dose of cefazolin prevents postoperative sepsis in high-risk biliary surgery. Can J Surg. 1984 Jan;27(1):44-7. PMID 6380693
- [Background] Lykkegaard Nielsen M, Moesgaard F, Justesen T, Scheibel JH, Lindenberg S. Wound sepsis after elective cholecystectomy. Restriction of prophylactic antibiotics to risk groups. Scand J Gastroenterol. 1981;16(7):937-40. doi: 10.3109/00365528109181826. PMID 7034165
- [Background] Landau O, Kott I, Deutsch AA, Stelman E, Reiss R. Multifactorial analysis of septic bile and septic complications in biliary surgery. World J Surg. 1992 Sep-Oct;16(5):962-4; discussion 964-5. doi: 10.1007/BF02067003. PMID 1462638
- [Background] Meijer WS. Antibiotic prophylaxis in biliary tract surgery--current practice in The Netherlands. Neth J Surg. 1990 Aug;42(4):96-100. PMID 2216008
- [Background] Havig O, Hertzberg J. [Effect of ampicillin, chloramphenicol and penicillin + streptomycin in the treatment of acute cholecystitis]. Tidsskr Nor Laegeforen. 1975 Feb 20;95(5):298-300. No abstract available. Norwegian. PMID 1118852
- [Background] Kune GA, Burdon JG. Are antibiotics necessary in acute cholecystitis? Med J Aust. 1975 Oct 18;2(16):627-30. PMID 1207539
- [Background] Groezinger KH. Prophylactic use of mezlocillin in acute cholecystitis. Chemioterapia. 1987 Jun;6(2 Suppl):590. No abstract available. PMID 3509507
- [Background] Muller EL, Pitt HA, Thompson JE Jr, Doty JE, Mann LL, Manchester B. Antibiotics in infections of the biliary tract. Surg Gynecol Obstet. 1987 Oct;165(4):285-92. PMID 3310282
- [Background] Friedlender J, Meyer P, Marti MC, Rohner A. Comparative study of ceftriaxone and cefoperazone in the treatment of acute cholecystitis. Chemotherapy. 1988;34 Suppl 1:30-3. doi: 10.1159/000238644. PMID 3246168
- [Background] Lau WY, Yuen WK, Chu KW, Chong KK, Li AK. Systemic antibiotic regimens for acute cholecystitis treated by early cholecystectomy. Aust N Z J Surg. 1990 Jul;60(7):539-43. doi: 10.1111/j.1445-2197.1990.tb07422.x. PMID 2113376
- [Background] Grant MD, Jones RC, Wilson SE, Bombeck CT, Flint LM, Jonasson O, Soroff HS, Stellato TA, Dougherty SH. Single dose cephalosporin prophylaxis in high-risk patients undergoing surgical treatment of the biliary tract. Surg Gynecol Obstet. 1992 May;174(5):347-54. PMID 1570609
- [Background] Krajden S, Yaman M, Fuksa M, Langer JC, Rowan J, Burul CJ, Wooster DL, Deitel M, Borowy ZJ, Smith LC, et al. Piperacillin versus cefazolin given perioperatively to high-risk patients who undergo open cholecystectomy: a double-blind, randomized trial. Can J Surg. 1993 Jun;36(3):245-50. PMID 8324671
- [Background] Chacon JP, Criscuolo PD, Kobata CM, Ferraro JR, Saad SS, Reis C. Prospective randomized comparison of pefloxacin and ampicillin plus gentamicin in the treatment of bacteriologically proven biliary tract infections. J Antimicrob Chemother. 1990 Oct;26 Suppl B:167-72. doi: 10.1093/jac/26.suppl_b.167. PMID 2258344
- [Background] Thompson JE Jr, Bennion RS, Roettger R, Lally KP, Hopkins JA, Wilson SE. Cefepime for infections of the biliary tract. Surg Gynecol Obstet. 1993;177 Suppl:30-4; discussion 35-40. PMID 8256189
- [Background] Mayumi T, Takada T, Kawarada Y, Nimura Y, Yoshida M, Sekimoto M, Miura F, Wada K, Hirota M, Yamashita Y, Nagino M, Tsuyuguchi T, Tanaka A, Gomi H, Pitt HA. Results of the Tokyo Consensus Meeting Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):114-21. doi: 10.1007/s00534-006-1163-8. Epub 2007 Jan 30. PMID 17252304
- [Background] Eskelinen M, Ikonen J, Lipponen P. Diagnostic approaches in acute cholecystitis; a prospective study of 1333 patients with acute abdominal pain. Theor Surg 1993;8:15-20
- [Background] Brewer BJ, Golden GT, Hitch DC, Rudolf LE, Wangensteen SL. Abdominal pain. An analysis of 1,000 consecutive cases in a University Hospital emergency room. Am J Surg. 1976 Feb;131(2):219-23. doi: 10.1016/0002-9610(76)90101-x. PMID 1251963
- [Background] Telfer S, Fenyo G, Holt PR, de Dombal FT. Acute abdominal pain in patients over 50 years of age. Scand J Gastroenterol Suppl. 1988;144:47-50. PMID 3165555
- [Background] [Acute abdominal pain. A prospective multicentric study (author's transl)]. Nouv Presse Med. 1981 Dec 19;10(46):3771-3. French. PMID 7033931
- [Background] Bjorvatn B. Cholecystitis--etiology and treatment--microbiological aspects. Scand J Gastroenterol Suppl. 1984;90:65-70. PMID 6610921
- [Background] Tokunaga Y, Nakayama N, Ishikawa Y, Nishitai R, Irie A, Kaganoi J, Ohsumi K, Higo T. Surgical risks of acute cholecystitis in elderly. Hepatogastroenterology. 1997 May-Jun;44(15):671-6. PMID 9222669
- [Background] Girard RM, Morin M. Open cholecystectomy: its morbidity and mortality as a reference standard. Can J Surg. 1993 Feb;36(1):75-80. PMID 8443723
- [Background] Addison NV, Finan PJ. Urgent and early cholecystectomy for acute gallbladder disease. Br J Surg. 1988 Feb;75(2):141-3. doi: 10.1002/bjs.1800750217. PMID 3349301
- [Background] Inoue T, Mishima Y. Postoperative acute cholecystitis: a collective review of 494 cases in Japan. Jpn J Surg. 1988 Jan;18(1):35-42. doi: 10.1007/BF02470844. PMID 3290556
- [Background] Savoca PE, Longo WE, Zucker KA, McMillen MM, Modlin IM. The increasing prevalence of acalculous cholecystitis in outpatients. Results of a 7-year study. Ann Surg. 1990 Apr;211(4):433-7. doi: 10.1097/00000658-199004000-00009. PMID 2322038
- [Background] Hafif A, Gutman M, Kaplan O, Winkler E, Rozin RR, Skornick Y. The management of acute cholecystitis in elderly patients. Am Surg. 1991 Oct;57(10):648-52. PMID 1928982
- [Background] Glenn F. Surgical management of acute cholecystitis in patients 65 years of age and older. Ann Surg. 1981 Jan;193(1):56-9. doi: 10.1097/00000658-198101000-00009. PMID 7458450
- [Background] Jarvinen HJ, Hastbacka J. Early cholecystectomy for acute cholecystitis: a prospective randomized study. Ann Surg. 1980 Apr;191(4):501-5. doi: 10.1097/00000658-198004000-00018. PMID 6445180
- [Background] van der Linden W, Sunzel H. Early versus delayed operation for acute cholecystitis. A controlled clinical trial. Am J Surg. 1970 Jul;120(1):7-13. doi: 10.1016/s0002-9610(70)80133-7. No abstract available. PMID 5426869
- [Background] Norrby S, Herlin P, Holmin T, Sjodahl R, Tagesson C. Early or delayed cholecystectomy in acute cholecystitis? A clinical trial. Br J Surg. 1983 Mar;70(3):163-5. doi: 10.1002/bjs.1800700309. No abstract available. PMID 6338991
- [Background] Siddiqui T, MacDonald A, Chong PS, Jenkins JT. Early versus delayed laparoscopic cholecystectomy for acute cholecystitis: a meta-analysis of randomized clinical trials. Am J Surg. 2008 Jan;195(1):40-7. doi: 10.1016/j.amjsurg.2007.03.004. PMID 18070735
- [Background] Kolla SB, Aggarwal S, Kumar A, Kumar R, Chumber S, Parshad R, Seenu V. Early versus delayed laparoscopic cholecystectomy for acute cholecystitis: a prospective randomized trial. Surg Endosc. 2004 Sep;18(9):1323-7. doi: 10.1007/s00464-003-9230-6. Epub 2004 Jul 7. PMID 15803229
- [Background] Lai PB, Kwong KH, Leung KL, Kwok SP, Chan AC, Chung SC, Lau WY. Randomized trial of early versus delayed laparoscopic cholecystectomy for acute cholecystitis. Br J Surg. 1998 Jun;85(6):764-7. doi: 10.1046/j.1365-2168.1998.00708.x. PMID 9667702
- [Background] Lo CM, Liu CL, Fan ST, Lai EC, Wong J. Prospective randomized study of early versus delayed laparoscopic cholecystectomy for acute cholecystitis. Ann Surg. 1998 Apr;227(4):461-7. doi: 10.1097/00000658-199804000-00001. PMID 9563529
- [Background] Johansson M, Thune A, Nelvin L, Stiernstam M, Westman B, Lundell L. Randomized clinical trial of open versus laparoscopic cholecystectomy in the treatment of acute cholecystitis. Br J Surg. 2005 Jan;92(1):44-9. doi: 10.1002/bjs.4836. PMID 15584058
- [Background] Kiviluoto T, Siren J, Luukkonen P, Kivilaakso E. Randomised trial of laparoscopic versus open cholecystectomy for acute and gangrenous cholecystitis. Lancet. 1998 Jan 31;351(9099):321-5. doi: 10.1016/S0140-6736(97)08447-X. PMID 9652612
- [Background] Alponat A, Kum CK, Koh BC, Rajnakova A, Goh PM. Predictive factors for conversion of laparoscopic cholecystectomy. World J Surg. 1997 Jul-Aug;21(6):629-33. doi: 10.1007/pl00012288. PMID 9230661
- [Background] Watson JF. The role of bacterial infection in acute cholecystitis: a prospective clinical study. Mil Med. 1969 Jun;134(6):416-26. No abstract available. PMID 4977359
- [Background] Calpena Rico R, Sanchez Llinares JR, Candela Polo F, Perez Vazquez MT, Vazquez Rojas JL, Diego Estevez M, Compan Rosique A, Medrano Heredia J. [Bacteriologic findings as a prognostic factor in the course of acute cholecystitis]. Rev Esp Enferm Apar Dig. 1989 Nov;76(5):465-70. Spanish. PMID 2616856
- [Background] Claesson B, Holmlund D, Matzsch T. Biliary microflora in acute cholecystitis and the clinical implications. Acta Chir Scand. 1984;150(3):229-37. PMID 6380177
- [Background] Csendes A, Burdiles P, Maluenda F, Diaz JC, Csendes P, Mitru N. Simultaneous bacteriologic assessment of bile from gallbladder and common bile duct in control subjects and patients with gallstones and common duct stones. Arch Surg. 1996 Apr;131(4):389-94. doi: 10.1001/archsurg.1996.01430160047008. PMID 8615724
- [Background] Jarvinen HJ. Biliary bacteremia at various stages of acute cholecystitis. Acta Chir Scand. 1980;146(6):427-30. PMID 7468075
- [Background] Linhares MM, Paiva V, Castelo Filho A, Granero LC, Pereira CA, Machado AM, Goldenberg A, Matos D. [Study of preoperative risk factors for bacteriobilia in patients with acute calculosis cholecystitis]. Rev Assoc Med Bras (1992). 2001 Jan-Mar;47(1):70-7. doi: 10.1590/s0104-42302001000100033. French. PMID 11340454
- [Background] Thompson JE Jr, Bennion RS, Doty JE, Muller EL, Pitt HA. Predictive factors for bactibilia in acute cholecystitis. Arch Surg. 1990 Feb;125(2):261-4. doi: 10.1001/archsurg.1990.01410140139024. PMID 2302066
- [Background] Pitt HA, Postier RG, Cameron JL. Consequences of preoperative cholangitis and its treatment on the outcome of operation for choledocholithiasis. Surgery. 1983 Sep;94(3):447-52. PMID 6612580
- [Background] Maluenda F, Csendes A, Burdiles P, Diaz J. Bacteriological study of choledochal bile in patients with common bile duct stones, with or without acute suppurative cholangitis. Hepatogastroenterology. 1989 Jun;36(3):132-5. PMID 2502489
- [Background] Kimura Y, Takada T, Kawarada Y, Nimura Y, Hirata K, Sekimoto M, Yoshida M, Mayumi T, Wada K, Miura F, Yasuda H, Yamashita Y, Nagino M, Hirota M, Tanaka A, Tsuyuguchi T, Strasberg SM, Gadacz TR. Definitions, pathophysiology, and epidemiology of acute cholangitis and cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):15-26. doi: 10.1007/s00534-006-1152-y. Epub 2007 Jan 30. PMID 17252293
- [Background] Hirota M, Takada T, Kawarada Y, Nimura Y, Miura F, Hirata K, Mayumi T, Yoshida M, Strasberg S, Pitt H, Gadacz TR, de Santibanes E, Gouma DJ, Solomkin JS, Belghiti J, Neuhaus H, Buchler MW, Fan ST, Ker CG, Padbury RT, Liau KH, Hilvano SC, Belli G, Windsor JA, Dervenis C. Diagnostic criteria and severity assessment of acute cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):78-82. doi: 10.1007/s00534-006-1159-4. Epub 2007 Jan 30. PMID 17252300
- [Background] Recommandations de la SFAR. Pour la pratique de l'antibioprophylaxie en chirurgie viscérale. J Chir1999;136:211-5.
- [Background] Juvonen T, Kiviniemi H, Niemela O, Kairaluoma MI. Diagnostic accuracy of ultrasonography and C reactive protein concentration in acute cholecystitis: a prospective clinical study. Eur J Surg. 1992 Jun-Jul;158(6-7):365-9. PMID 1356470
- [Background] Hakansson K, Leander P, Ekberg O, Hakansson HO. MR imaging in clinically suspected acute cholecystitis. A comparison with ultrasonography. Acta Radiol. 2000 Jul;41(4):322-8. doi: 10.1080/028418500127345587. PMID 10937751
- [Background] De Vargas Macciucca M, Lanciotti S, De Cicco ML, Coniglio M, Gualdi GF. Ultrasonographic and spiral CT evaluation of simple and complicated acute cholecystitis: diagnostic protocol assessment based on personal experience and review of the literature. Radiol Med. 2006 Mar;111(2):167-80. doi: 10.1007/s11547-006-0018-3. English, Italian. PMID 16671375
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Weigand K, Koninger J, Encke J, Buchler MW, Stremmel W, Gutt CN. Acute cholecystitis - early laparoskopic surgery versus antibiotic therapy and delayed elective cholecystectomy: ACDC-study. Trials. 2007 Oct 4;8:29. doi: 10.1186/1745-6215-8-29. PMID 17916243
- [Result] Fuks D, Duhaut P, Mauvais F, Pocard M, Haccart V, Paquet JC, Millat B, Msika S, Sielezneff I, Scotte M, Chatelain D, Regimbeau JM. A retrospective comparison of older and younger adults undergoing early laparoscopic cholecystectomy for mild to moderate calculous cholecystitis. J Am Geriatr Soc. 2015 May;63(5):1010-6. doi: 10.1111/jgs.13330. Epub 2015 May 6. PMID 25946647
- [Derived] Regimbeau JM, Fuks D, Pautrat K, Mauvais F, Haccart V, Msika S, Mathonnet M, Scotte M, Paquet JC, Vons C, Sielezneff I, Millat B, Chiche L, Dupont H, Duhaut P, Cosse C, Diouf M, Pocard M; FRENCH Study Group. Effect of postoperative antibiotic administration on postoperative infection following cholecystectomy for acute calculous cholecystitis: a randomized clinical trial. JAMA. 2014 Jul;312(2):145-54. doi: 10.1001/jama.2014.7586. PMID 25005651